CLINICAL TRIAL: NCT04421625
Title: Patients and Health Staff of Cancer Centres During the Covid-19 Pandemic: Constitution of a Biological Collection Linked to a Prospective, Multicenter Cohort Study
Brief Title: Patients and Health Staff of Cancer Centres During the Covid-19 Pandemic
Acronym: PAPESCO-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ICO-2020-16
Record Dates: First submitted 2020-05-18; First posted 2020-06-09 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: COVID-19; Cancer patients; Health staff
MeSH Terms: conditions — COVID-19 | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic test for SARS-Cov2 for patients and health staff (Experimental): * Blood test (rapid serology (immediate analysis), ELISA serology (differed analysis on frozen sample), genotyping of FCGR2A and FCGR3A gens)
  * Nasal swab test (only if the patient has symptoms)
  * Questionnaires
  Interventions: Diagnostic Test: Diagnostic test for SARS-Cov2 for patients and health staff

INTERVENTIONS:
Diagnostic Test: Diagnostic test for SARS-Cov2 for patients and health staff — Diagnostic test for SARS-CoV2 :
  * Blood test to analyse the IgG and IgM with an immediate qualitative analysis (serological test) and a differed quantitative analysis (ELISA test)
  * Results of nasal swab that will allow extracting the RNA and realizing a RT-PCR (only if the participants present symptoms). It will be obtained by standard local laboratories.
  * Questionnaires (based on serology, clinic, economy (socio-demographic and lifestyle questionnaire) and epidemiology)

SUMMARY:
The Covid-19 has, in a few weeks, made the world tremble: the number of deaths (mainly elderly and / or co-morbid) continues to increase, the confinement causes the collapsing of the economy and the decline of relationships inter-human. The data are too fragmented and the disease too recent to know its repercussions on the 3 million French people who have or have had cancer. The investigators would like, in 3 populations: * patients in treatment, * or in follow-up and * health personnel, to constitute a large prospective and longitudinal database of data: i / serological: humoral response, test performance, monitoring of serum immunoglobulin levels , reinfection threshold,…; ii / clinical: incidence, severity, mortality and their favorable factors impact of cancer treatment on Covid-19 infection and modification of the quality of oncological care in the context. In parallel, on a more limited sample of establishments, it will be : * appreciate the economic and functional repercussions, * will try to find out about the infection modalities in patients and health personnel and * will appreciate the levels of anxiety and depression to which health staff are subject.

DETAILED DESCRIPTION:
The participation of the study will be offered to each patient when they will come to the centre (by oncologist, radiotherapist, surgeon, ...). For the health staff, the information can be delivered through different channels (posting, mail, mail, intranet...). This will make the informed consent available to all staff. Participation will be voluntary: staff who have read the information note and wish to participate in the study will have to register on the "PAPESCO-01" screening schedule, during which they will sign their consent with the occupational physician (or anyone delegated by occupational medicine), then have their first sample and complete the various questionnaires.

The screening of the patients and of the health staff will be done by 2 or 3 techniques depending of the results. The first technic is a blood test done at M0 (inclusion), M3, M6, M9 and M12 and on demand in case of Covid-19 symptoms (rapid serology (immediate analysis), ELISA serology (differed analysis on frozen sample), genotyping of FCGR2A and FCGR3A gens (only at M0)). The second technic nasal swab test (RT-PCR) is done only in case of symptoms (whatever the result of the minute test is) for the hospitalized patients. The results of the tests realised in town will be get back through the questionnaires. The third technic is the questionnaires to the patients and the health staff.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Population in Cancer centres responding to one of these 3 definitions: patients having a treatment in process, patients under surveillance ( having completed their treatment for more than a year), health staff.
* Subjects who may or may not have had an infection compatible or proven with a Covid-19 infection.
* Information to the participants and signature of the informed consent.
* Subject affiliated with a social insurance

Exclusion Criteria:

* Refusal of consent
* Patients who are unable to consent or have a psychiatric history
* Inability to submit to the medical follow-up of the study for geographical, social or psychological reasons
* Person under guardianship or protection of vulnerable adults
* Person deprived of liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1102 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Bigot, MD, Study Director — Institut de Cancérologie de l'Ouest
Locations (3):
- France (3):
  - Institut de Cancerologie de l'Ouest, Angers
  - Centre Jean Perrin, Clermont-Ferrand
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic Test for SARS-Cov2 for Health Staff; Diagnostic Test for SARS-Cov2 for Patients: * Blood test (rapid serology (immediate analysis), ELISA serology (differed analysis on frozen sample), genotyping of FCGR2A and FCGR3A gens)
  * Nasal swab test (only if the patient has symptoms)
  * Questionnaires
  Diagnostic test for SARS-Cov2 for patients and health staff: Diagnostic test for SARS-CoV2 :
  * Blood test to analyse the IgG and IgM with an immediate qualitative analysis (serological test) and a differed quantitative analysis (ELISA test)
  * Results of nasal swab that will allow extracting the RNA and realizing a RT-PCR (only if the participants present symptoms). It will be obtained by standard local laboratories.
  * Questionnaires (based on serology, clinic, economy (socio-demographic and lifestyle questionnaire) and epidemiology)
Period: Overall Study
Arm/Group | Diagnostic Test for SARS-Cov2 for Health Staff | Diagnostic Test for SARS-Cov2 for Patients
Started | 579 | 523
Completed | 579 | 523
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diagnostic Test for SARS-Cov2 for Health Staff | Diagnostic Test for SARS-Cov2 for Patients | Total
Number analyzed (Participants) | 579 | 523 | 1102
Age, Continuous [Median (Full Range); unit: Years] | 40 [19 to 64] | 62 [27 to 89] | 51 [19 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 482 | 377 | 859
  Male | 97 | 146 | 243
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 579 | 523 | 1102

OUTCOME MEASURES:

1. Primary Outcome: Number and Severity of Confirmed COVID-19 Infections Among Cancer Centre Staff and Patients at 12 Months
Description: COVID-19 severity will be assessed using the World Health Organization Clinical Progression Scale, which ranges from 0 (uninfected) to 10 (death). Higher scores indicate worse clinical status. COVID-19 infection will be confirmed by PCR or antigen test. Data on symptoms and progression will be collected through a COVID-19 clinical signs follow-up questionnaire and verified by medical records. The outcome will report both the number of participants with confirmed infection and the distribution of severity scores across the scale.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic test for SARS-Cov2 for health staff | Diagnostic test for SARS-Cov2 for patients
Number analyzed (Participants) | 579 | 523
Participants | 55 | 36

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Diagnostic Test for SARS-Cov2 for Patients | Diagnostic Test for SARS-Cov2 for Health Staff
All-Cause Mortality (participants affected / at risk) | 0/523 | 0/579
Serious Adverse Events (participants affected / at risk) | 0/523 | 0/579
Other Adverse Events (participants affected / at risk) | 0/523 | 0/579

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT04421625/Prot_000.pdf